CLINICAL TRIAL: NCT04487392
Title: Photobiomodulation Effect on Vulvovaginal Atrophy in Postmenopausal Women: Randomized and Controlled Trial.
Brief Title: Photobiomodulation Effect on Vulvovaginal Atrophy in Postmenopausal Women.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The student do not start the study
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, INVESTIGATOR, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEDATROPHY
Record Dates: First submitted 2020-07-24; First posted 2020-07-27 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2020-07

CONDITIONS: Vulvovaginal Atrophy
Keywords: genitourinary syndrome; LED; light emitting diode; vulvovaginal atrophy; menopause; climacteric; photobiomodulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estrogen vaginal cream group (group A) (Active Comparator): 22 participants will be included in this group. The participants selected for group A will be provided with estriol 0.01% vaginal cream, which should be applied at home.
  Interventions: Drug: Estrogen vaginal cream group (group A)
- Photobiomodutation group (group B) (Experimental): 22 participants will be included in this group. The participants selected for group B will be undergo photobiomodulation with red LED.
  Interventions: Radiation: Photobiomodutation group (group B)

INTERVENTIONS:
Drug: Estrogen vaginal cream group (group A) — The participants selected for group A will be provided with estriol 0.01% vaginal cream, which should be applied at home: 1 intravaginal applicator at night, daily for 2 weeks, followed by 2 times a week, on alternate days (Monday - Thursday) for another 2 weeks.
  Arms: Estrogen vaginal cream group (group A)
Radiation: Photobiomodutation group (group B) — The participants selected for group B will be undergo photobiomodulation with red LED. With the participant in the lithotomy position, the speculum will be introduced into the vaginal canal and a vaginal wash with 0.9% saline will be performed to remove secretions. Afterwards, the speculum will be removed and the device with a red LED inserted up to about 6 cm from the introitus. A non-lubricated condom will be used in the LED device for patient protection. Sessions will take place once a week for 4 weeks.
  Arms: Photobiomodutation group (group B)

SUMMARY:
Menopause is a physiological event and is defined as the loss of ovarian follicular activity, with consequent permanent cessation of menstrual cycles. Its diagnosis is made retrospectively after 12 months of amenorrhea, with no pathological cause involved. This period is marked by several changes in the female organism, mainly the genitourinary syndrome (GUS), which is a collection of signs and symptoms resulting from the state of hypoestrogenism. Almost half of postmenopausal women will experience symptoms of GUS, with vaginal dryness being the most prevalent, followed by dyspareunia and vulvovaginal irritation. The aim of the study is to evaluate the effect of photobiomodulation with red LED (ligth emitting diode) on the symptoms of vulvovaginal atrophy in postmenopausal women. A randomized and controlled clinical trial will be developed, which will include postmenopausal women with signs and symptoms of vulvovaginal atrophy. Participants will be allocated into two groups: those who will undergo photobiomodulation with intravaginal LED, and those who will receive vaginal cream with estriol. Objective and subjective improvement of atrophy will be assessed using the Vaginal Health Index and the visual analog scale, respectively. Vaginal pH, cell maturation index and changes in sexual function through the Female Sexual Function Index questionnaire will also be assessed. The variables will be analyzed at the time of admission, in one and three months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women (amenorrhea for less than 12 months);
* presence one or more symptoms of vulvovaginal atrophy (dyspareunia, dryness, irritation and vaginal burning);
* Vaginal Heath Index ≤ 15 (signs of atrophy);
* normal cytopathology of uterine cervix in the last year.

Exclusion Criteria:

* previous or current history of gynecological neoplasia;
* who used hormonal or non-hormonal treatment for vulvovaginal symptoms of menopause;
* current or recent genitourinary lesions or infectious processes in the genitourinary tract (last month);
* current or recent (last month) systemic treatment with antifungals, antibiotics or corticosteroids;
* presence of genital prolapse;
* presence of contraindications to the use of vaginal estrogen (current, previous or suspected diagnosis of breast cancer, malignant estrogen-dependent tumors, uninvestigated uterine bleeding, untreated endometrial hyperplasia, deep venous thrombosis and current or previous pulmonary thromboembolism, known thrombophilia, recent or active arterial disease, acute liver disease, porphyria, use of drugs that may interact with estriol and hypersensitivity to the components of the vaginal cream formula).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective assessment of improvement in vulvovaginal atrophy symptoms. | 6 months
  Vaginal Health Index: an objective assessment will be performed using the parameters of the Vaginal Health Index, in which elasticity, fluid volume, pH, epithelial integrity and moisture are evaluated. Each aspect evaluated receives a score, which varies from 1 to 5. The score can vary from 5 to 25, being considered a diagnosis of vulvovaginal atrophy when the values are less than or equal to 15. This evaluation will be performed by a qualified gynecologist during the exam physicist.
Subjetive assessment of improvement in vulvovaginal atrophy symptoms. | 6 months
  Visual Analog scale: the assessment of vulvovaginal atrophy symptoms will be made using the visual analog scale. The patient will receive a ruler with markings from 0 to 10, one end of which indicates complete absence of symptoms and the other indicates the worst possible symptom. This assessment will be applied to each of the symptoms: dyspareunia, dryness, irritation.

SECONDARY OUTCOMES:
Vaginal pH | 6 months
  The evaluation of the vaginal pH will be performed through the pH indicator strip, which when inserted in the middle third of the vagina in contact with the mucosa, has the color of the strip changed.
Female Sexual Function Index | 6 months
  The quality of the participants' sexual activity will be assessed through the questionnaire validated for the Portuguese "Female Sexual Function Index". This questionnaire is a brief and self-applied instrument that assesses the female sexual response in the last four weeks in relation to sexual desire, vaginal lubrication, orgasm, sexual satisfaction and pain.
Vaginal Cell Maturation Index | 6 months
  Also known as Frost Index, whose aim is to assess the hormonal influence in women by counting the epithelial cells of the vagina. The frequencies of parabasal, intermediate and superficial cells are evaluated. For this, a scraping of the lateral wall of the vagina is performed with a spatula, in order to obtain vaginal cells for cytology. The cells will be fixed on a slide and later colored with HE (Hematoxylin-Eosin) for analysis and counting.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davis SR, Lambrinoudaki I, Lumsden M, Mishra GD, Pal L, Rees M, Santoro N, Simoncini T. Menopause. Nat Rev Dis Primers. 2015 Apr 23;1:15004. doi: 10.1038/nrdp.2015.4. PMID 27188659
- [Background] Schoenaker DA, Jackson CA, Rowlands JV, Mishra GD. Socioeconomic position, lifestyle factors and age at natural menopause: a systematic review and meta-analyses of studies across six continents. Int J Epidemiol. 2014 Oct;43(5):1542-62. doi: 10.1093/ije/dyu094. Epub 2014 Apr 26. PMID 24771324
- [Background] Takahashi TA, Johnson KM. Menopause. Med Clin North Am. 2015 May;99(3):521-34. doi: 10.1016/j.mcna.2015.01.006. PMID 25841598
- [Background] Gandhi J, Chen A, Dagur G, Suh Y, Smith N, Cali B, Khan SA. Genitourinary syndrome of menopause: an overview of clinical manifestations, pathophysiology, etiology, evaluation, and management. Am J Obstet Gynecol. 2016 Dec;215(6):704-711. doi: 10.1016/j.ajog.2016.07.045. Epub 2016 Jul 26. PMID 27472999
- [Background] Kingsberg SA, Wysocki S, Magnus L, Krychman ML. Vulvar and vaginal atrophy in postmenopausal women: findings from the REVIVE (REal Women's VIews of Treatment Options for Menopausal Vaginal ChangEs) survey. J Sex Med. 2013 Jul;10(7):1790-9. doi: 10.1111/jsm.12190. Epub 2013 May 16. PMID 23679050
- [Background] Pacagnella Rde C, Martinez EZ, Vieira EM. [Construct validity of a Portuguese version of the Female Sexual Function Index]. Cad Saude Publica. 2009 Nov;25(11):2333-44. doi: 10.1590/s0102-311x2009001100004. Portuguese. PMID 19936472